CLINICAL TRIAL: NCT00468962
Title: The Effct of Chitooligosaccharide on Immune Function in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eulji University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 07-05
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2007-05-03 (Estimated); Status verified 2007-05

CONDITIONS: Immunity
MeSH Terms: interventions — Functional Food

INTERVENTIONS:
Drug: FACOS (functional food)

SUMMARY:
Functional properties of chitooligosaccharides have been studied for antitumor activity, immunostimulating effects, antimicrobial activity, free radical scavening activity, adn angiotensin I converting enzyme inhibitory activity. Recent in vitro, and in vivo toxicity and absorbability studies have demonstrated that chitooligosaccharides have high absorbability and are essentially non-toxic. In the present study, we prepared a chitooligosaccharide with high absorbability and evaluated its effects on activation of immune function and cardiovascular funciton(lipid, atrial stiffness, etc) in healthy adults.

This study was a 8-week, randomized, double-blind clinical trial. The 30 volunteers were divided into a control group(n=10), half dose chitooligosaccaride(FACOSTM) intake group(n=10), and full dose FACOS intake group(n=10). Peripheral blood mononuclear cells(PBMCs) were isolated and cultured in 12 well plate for 48 hours. Cytokine production by PBMCs pre- and postintervention were measured simultaneously after stimulation with lipopolysaccaride.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults(the ages between 20~50 year)

Exclusion Criteria:

* food allergy and allergy skin disease
* severe liver and kidney disease
* pregnant, lactating women
* cancer, stroke, etc.

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Jeong Choi, MD, Ph.D, Principal Investigator — Eulji University Hospital